CLINICAL TRIAL: NCT05334459
Title: Preoperative Radiotherapy and Systemic Therapy Following Surgery in 'de Novo' Metastatic Breast Cancer (Protocol MF22-01; Intervention Systemic Treatment METastasis-ISTMET)
Brief Title: Preoperative Radiotherapy and Systemic Therapy Following Surgery in 'de Novo' Metastatic Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Ankara Oncology Research and Training Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ISTMET-BHWGI2022-1
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Metastatic Breast Cancer
Keywords: breast cancer, metastasis, radiotherapy, primer surgery
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intervention: Operable, postmenopausal ER/PR positive and Her2 neu (-), oligometastatic dnMBC patients
  * Primary tumor biopsy, Metastatic site biopsy (Bone, liver, etc)
    o ER / PR /Her2 /Ki67 study
  * Collection of CTC.
  * Radiotherapy (RT) to the primary breast tumor (Hypo fractionated)
  * All patients will receive the standard of care treatment with CDK4/6 inhibitor + AI for 6 months (at least 26 weeks).
    o Denosumab, Biphosphonate for bone metastasis
  * RT to metastatic side (if visible). Continue Systemic therapy
  * 12 months, patients will have LRT surgery (BCS/mastectomy + LN evaluation; SLNB+ALND) + RT (based on the institutional practice). Collect CTC and ER/PR/Her 2 in the final specimen
  * ST will be continued until progression and/or unmanageable toxicity.
  * Radiologic evaluation every 3-6-month based on institutional practice.
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — Oligometastatic disease (defined here as 5 or fewer sites of metastatic disease involving 3 or fewer organ systems)
  * Primary tumor biopsy, Metastatic site biopsy (Bone, liver, etc) (if there is, based on institutional practice)
    o ER / PR /Her2 /Ki67 study)
  * Collection of CTC.
  * Radiotherapy (RT) to the primary breast tumor (Hypo fractionated)
  * All patients will receive the standard of care treatment with CDK4/6 inhibitor + AI for 6 months (at least 26 weeks).
    o Denosumab, Biphosphonate for bone metastasis
  * RT to metastatic side (if visible). Continue Systemic therapy
  * 12 months, patients will have LRT surgery (BCS/mastectomy + LN evaluation; SLNB+ALND) + RT (based on the institutional practice). Collect CTC and ER/PR/Her 2 in the final specimen
  * ST will be continued until progression and/or unmanageable toxicity.
  * Radiologic evaluation every 3-6-month based on institutional practice.

SUMMARY:
Locoregional (LRT) of the primary tumor in de-novo metastatic breast cancer (dnMBC) is no longer only a surgical challenge, but more the final decision of a multidisciplinary tumor board including medical oncologists, radiation oncologists and surgical oncologists. It is no longer only a question of locoregional control but rather a wider issue of improving overall survival (OS), due to the possible biological link between primary tumor and metastases. A multimodal approach, including LRT with curative intent should be considered for selected dnMBC patients, especially for the subset of bone-only metastatic ones.

DETAILED DESCRIPTION:
Five to eight percent of breast cancer (BC) patients present with distant metastasis at diagnosis which is known as 'de novo' metastatic breast cancer (dnMBC). These patients represent up to 25% of all MBC patients and tend to have more favorable prognosis than those who relapse during follow-up. Recent data showed that approximately 40% of dnMBC patients undergo locoregional treatment (LRT). Most of the retrospective series over the past two decades showed that LRT not only controls locoregional progression, but also contributes to overall survival (OS), moreover meta-analyses suggest that surgical resection of the primary tumor may improve OS with a hazard ratio (HR) of around 0.60. MF07-01 study, one of the first clinical randomized trials, showed that the patients with diagnosis of dnMBC undergoing LRT followed by systemic therapy had an additional 14% OS benefit by the end of the 10-year follow-up when compared with patients who received only systemic therapy.

Patient-related factors (i.e. age, comorbidities), metastatic burden (i.e. site and number of metastases) and more prominently tumor biology are major factors for therapeutic decisions in dnMBC. Metastatic sites differ according to the intrinsic BC subtypes. Bone and lymph nodes are more common sites for metastasis in hormone receptor (ER, PR) positive BC patients whereas visceral and brain metastasis is more common in Her2 positive & triple negative BC. Tailored therapy, such as targeted therapy & immunotherapy is based on IHC profile, genetic & molecular features in intrinsic subtypes (i.e. luminal A-like, luminal B-like Her2 negative, luminal B-like Her2 positive, Her2 positive nonluminal & basal-like breast cancer). Tailored therapy contributes to survival outcomes.

Aromatase inhibitors (AI: anastrozole, letrozole, exemestane) with cyclin dependent kinase 4/6 inhibitors (CDKi: ribociclib, palbociclib, abemaciclib) are standard of care as first line setting in postmenopausal metastatic Her2 negative luminal-like breast cancer (mHN-LBC) patients. In the last decade, first line AI/CDKi combination has been shown to increase progression free survival (PFS) and objective response rates (ORR). Recently, updated OS outcomes with a median follow-up of more than 6.5 years has been presented at ESMO congress in September 2021. It has been reported that first line ribociclib and letrozole combination has been shown to have significant OS advantage over letrozole in mHN- 2 LBC. So, AI/CDKi combination as first line systemic treatment in postmenopausal mHN-LBC significantly decreases both progression and mortality rates. In Turkey, ribociclib and palbociclib are available options as CDKi. Therefore, AI/CDKi (ribociclib/palbociclib) combination is also preferred as first line setting for postmenopausal mHN-LBC in our country.

Hormone receptor (ER, PR) and Her2 positivity might differ for primary & metastatic sites in BC, especially in relapsed patients. Discordance (i.e 'positivity conversion to negativity' or 'negativity conversion to positivity') rates are reported as 10-30% for ER, 20-50% for PR and 10-15% for Her2 in relapsed MBC, but data is limited for dnMBC. It has been reported that total discordance rate as 27% for ER / PR and/or Her2 between primary tumor and metastatic sites in MBC. It was 14.26% for ER/PR & 7.8% for Her2 status, respectively. They evaluated 16703 MBC patients in a large scale real-life multicenter French ESME cohort. In this cohort, 2169 patients had biopsy from both primary tumor and metastatic site within 6 months of MBC diagnosis, only 10% (n:1677) had optimal biopsy material for ER/PR & Her2 discordance evaluation. Taking into account these high discordance rates, synchronous biopsy from primary tumor and metastatic sites should be preferred in prospective clinical trial designs in dnMBC. However, it might not be so easy and pragmatic in daily practice.

Moreover, radiotherapy (RT) techniques have considerably improved, allowing for the radiation dose to conform more precisely to the three-dimensional shape of the tumor, thus enabling much higher radiation doses and better tumor control with less toxicity.

Observational studies showed that bone was the most common site of metastasis (around 45% of patients) and up to 30% of patients were diagnosed with bone-only metastases. For oligometastatic disease, some retrospective and prospective series demonstrated that local treatment of all metastases, when feasible, was significantly associated with prolonged survival. Patients with oligometastatic bone-only MBC treated with stereotactic radiotherapy had better clinical outcomes than those who had metastasis at other sites. It has been reported that local breast surgery was associated with better survival outcomes for the patients with only one metastatic site involvement (i.e. bone, liver or lung), but not for brain-only metastasis when they stratified the patients according to the distant metastatic sites. Our study group (BOMET trial) demonstrated that LRT prolonged survival and decreased locoregional recurrence in a prospectively maintained registry study with a median follow-up of 3 years, previously. Timing of primary breast surgery either at diagnosis or after systemic treatment provided a survival benefit similar to systemic therapy alone in bone-only dnMBC patients. Two ongoing prospective phase III trials (NCT02089100, NCT02364557) are evaluating the role of metastases local ablation (Stereotactic Body Radiation therapy (SBRT) or surgery) with curative intent in oligometastatic breast cancer.

In conclusion, LRT of the primary tumor in dnMBC is no longer only a surgical challenge, but more the final decision of a multidisciplinary tumor board including medical oncologists, radiation oncologists and surgical oncologists. It is no longer only a question of locoregional control but rather a wider issue of improving OS, due to the possible biological link between primary tumor and metastases. A multimodal approach, including LRT with curative intent should be considered for selected dnMBC patients, especially for the subset of bone-only metastatic ones.

ELIGIBILITY:
Inclusion Criteria:

* Primary breast tumor amenable for complete surgical resection, patients in good physical condition for receiving protocol driven locoregional and systemic treatments and receiving radiotherapy.

Exclusion Criteria:

* Primary tumor not amenable for complete resection; primary tumor with extended infection, bleeding, or necrosis; patients with poor physical condition which prevents the patient from receiving protocol driven locoregional and systemic treatment; synchronous primary cancer at the contralateral breast; clinically involved contralateral axillary nodes; patients not suitable for adequate follow-up, and failure to give informed consent. Pregnancy and lactation.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Operable, postmenopausal ER/PR positive and Her2 neu (-), oligometastatic dnMBC patients.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years follow-up
  Phase I study to evaluate feasibility (overall and diseas free survival) of this curative intent treatment approach to patients presenting with dnMBC with oligometastatic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Serdar Ozbas, Prof, Principal Investigator — Endocrine and Breast Surgeon-Ankara; Atilla Soran, Prof, Study Chair — Magee-Womens Hospital,University of Pittsburgh Medical Center
Locations (1):
- Lutfi Dogan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soran A, Ozmen V, Ozbas S, Karanlik H, Muslumanoglu M, Igci A, Canturk NZ, Utkan Z, Evrensel T, Sezgin E; MF07-01 Study Group. Primary Surgery with Systemic Therapy in Patients with de Novo Stage IV Breast Cancer: 10-year Follow-up; Protocol MF07-01 Randomized Clinical Trial. J Am Coll Surg. 2021 Dec;233(6):742-751.e5. doi: 10.1016/j.jamcollsurg.2021.08.686. Epub 2021 Sep 13. PMID 34530124
- [Background] Lee SJ, Park S, Ahn HK, Yi JH, Cho EY, Sun JM, Lee JE, Nam SJ, Yang JH, Park YH, Ahn JS, Im YH. Implications of bone-only metastases in breast cancer: favorable preference with excellent outcomes of hormone receptor positive breast cancer. Cancer Res Treat. 2011 Jun;43(2):89-95. doi: 10.4143/crt.2011.43.2.89. Epub 2011 Jun 30. PMID 21811424
- [Background] Sledge GW Jr, Toi M, Neven P, Sohn J, Inoue K, Pivot X, Burdaeva O, Okera M, Masuda N, Kaufman PA, Koh H, Grischke EM, Conte P, Lu Y, Barriga S, Hurt K, Frenzel M, Johnston S, Llombart-Cussac A. The Effect of Abemaciclib Plus Fulvestrant on Overall Survival in Hormone Receptor-Positive, ERBB2-Negative Breast Cancer That Progressed on Endocrine Therapy-MONARCH 2: A Randomized Clinical Trial. JAMA Oncol. 2020 Jan 1;6(1):116-124. doi: 10.1001/jamaoncol.2019.4782. PMID 31563959
- [Background] Onderdonk BE, Gutiontov SI, Chmura SJ. The Evolution (and Future) of Stereotactic Body Radiotherapy in the Treatment of Oligometastatic Disease. Hematol Oncol Clin North Am. 2020 Feb;34(1):307-320. doi: 10.1016/j.hoc.2019.09.003. Epub 2019 Oct 28. PMID 31739951
- [Background] Wang K, Shi Y, Li ZY, Xiao YL, Li J, Zhang X, Li HY. Metastatic pattern discriminates survival benefit of primary surgery for de novo stage IV breast cancer: A real-world observational study. Eur J Surg Oncol. 2019 Aug;45(8):1364-1372. doi: 10.1016/j.ejso.2019.02.013. Epub 2019 Feb 19. PMID 30837102
- [Background] Trovo M, Furlan C, Polesel J, Fiorica F, Arcangeli S, Giaj-Levra N, Alongi F, Del Conte A, Militello L, Muraro E, Martorelli D, Spazzapan S, Berretta M. Radical radiation therapy for oligometastatic breast cancer: Results of a prospective phase II trial. Radiother Oncol. 2018 Jan;126(1):177-180. doi: 10.1016/j.radonc.2017.08.032. Epub 2017 Sep 21. PMID 28943046
- [Background] Milano MT, Katz AW, Zhang H, Huggins CF, Aujla KS, Okunieff P. Oligometastatic breast cancer treated with hypofractionated stereotactic radiotherapy: Some patients survive longer than a decade. Radiother Oncol. 2019 Feb;131:45-51. doi: 10.1016/j.radonc.2018.11.022. Epub 2018 Dec 28. PMID 30773186
- [Background] Soran A, Dogan L, Isik A, Ozbas S, Trabulus DC, Demirci U, Karanlik H, Soyder A, Dag A, Bilici A, Dogan M, Koksal H, Sendur MAN, Gulcelik MA, Maralcan G, Cabioglu N, Yeniay L, Utkan Z, Simsek T, Karadurmus N, Daglar G, Yildiz B, Uras C, Tukenmez M, Yildirim A, Kutun S, Ozaslan C, Karaman N, Akcay MN, Toktas O, Sezgin E. The Effect of Primary Surgery in Patients with De Novo Stage IV Breast Cancer with Bone Metastasis Only (Protocol BOMET MF 14-01): A Multi-Center, Prospective Registry Study. Ann Surg Oncol. 2021 Sep;28(9):5048-5057. doi: 10.1245/s10434-021-09621-8. Epub 2021 Feb 2. PMID 33532878